CLINICAL TRIAL: NCT05597644
Title: Role of Uterine Artery Angioembolization in Management of Uterine Adenomyosis.
Brief Title: Role of Uterine Artery Embolization in Adenomyosis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moustafa Tarek Khalaf Al-Hussaini, Specialist, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAE in adenomyosis
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-05

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Intervention Model Description: Angioembolization of uterine artery by PVA particles
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- females with adenomyosis (Experimental)
  Interventions: Procedure: Trans-arterial uterine artery embolization

INTERVENTIONS:
Procedure: Trans-arterial uterine artery embolization — transarterial angioembolization of uterine artery

SUMMARY:
Management of symptomatizing women diagnosed with uterine adenomyosis, by uterine artery angioembolization as a minimally invasive replacement for hysterectomy. This is followed by assessment of the symptoms and MRI of the pelvis after 3 months.

DETAILED DESCRIPTION:
Adenomyosis is defined by the abnormal location of endometrial tissue within the myometrium associated with hypertrophy or hyperplasia of the myometrial stroma. Although pathogenesis and etiology of adenomyosis remain unknown, two main theories have been proposed: invagination of the endometrial basal layer and metaplasia of embryonic stem cells. Despite the absence of specific (pathognomonic) diagnostic features for uterine adenomyosis, typical symptoms include menorrhagia, chronic pelvic pain, and dysmenorrhea.

For more than a century, diagnosis was dependent on histopathologic examination of post-hysterectomy specimens till the introduction of noninvasive ultrasound and MR techniques. Since then, several studies have illustrated high sensitivities and specificities for both two-dimensional transvaginal sonography (TVS) and magnetic resonance imaging (MRI). Current treatment options for symptomatic adenomyosis include hysterectomy, medication, conservative surgery, or minimally invasive techniques including uterine artery embolization. To date, hysterectomy remains the definitive treatment. This is mainly due to difficult diagnosis, the diffuse nature of the disease, and little evidence-based literature needed to standardize treatments. This consequently results in a management dilemma, particularly in symptomatic patients who wish to preserve their uterus.

Uterine artery embolization is the use of transarterial catheters aiming to induce more than 34% necrosis within adenomyotic tissues. Vascular access is gained through a femoral or radial artery puncture using 4-6-French (F) arterial sheath for femoral and 4-F sheath for radial access. Under fluoroscopic guidance, aortography is followed by selective and super selective arteriography using 4-5-F catheters for the internal iliac and 2-3-F microcatheters for the uterine artery and its branches respectively. Embolization is usually performed using variable-sized permanent particulate agents.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatizing women (pelvic pain and/or bleeding) between ages 30-50 who are not keen on hysterectomy.

Exclusion Criteria:

* Women who desire further child bearing (not completed their family yet).
* Impaired coagulation profile.
* Hypersensitivity to intravenous contrast media.
* Decompensated congestive heart failure.
* Hypertensive crisis.
* Stroke or CVA.
* Renal failure.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
uterine artery embolization in management of adenomyosis | baseline
  study the effect of embolization on symptoms and imaging findings

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Mansour, Assistant Professor, Study Director — Assiut University; Abd ElKareem Hasan, Professor, Study Chair — Assiut University